CLINICAL TRIAL: NCT05574010
Title: A Phase 1B Open-label/Phase 2 Double-blind Placebo- Controlled Study for Pharmacodynamic (PD) Activity, Pharmacokinetics (PK), Safety, and Tolerability of KAN-101 In Patients With Celiac Disease (CeD)
Brief Title: A Study of Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of KAN-101 in Celiac Disease (ACeD-it)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Kanyos Bio, Inc., a wholly-owned subsidiary of Anokion SA (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Anokion SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KAN-101-02
Record Dates: First submitted 2022-10-07; First posted 2022-10-10 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Celiac Disease
Keywords: celiac disease; HLA-DQ2.5; gluten free diet
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: Part A: This part of the study is an open label with up to 6 participants in each dose cohort. There will be 2 dose cohorts.
  Part B and Part C: These parts of the study have a randomized, double- blinded, placebo-controlled, parallel study design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part A is open label Part B and Part C are a double-blinded study. Study participants and their caregivers, investigators and other site staff, and sponsor staff involved in the study team will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 in Part A (Experimental): All eligible Part A participants will receive 3 intravenous (IV) infusions of KAN-101 Dose 1
  Interventions: Drug: Cohort 1 in Part A
- Cohort 2 in Part A (Experimental): All eligible Part A participants will receive 3 intravenous (IV) infusions of KAN-101 Dose 2
  Interventions: Drug: Cohort 2 in Part A
- Group 1 in Part B and Part C (Placebo Comparator): All eligible Part B and Part C participants will receive 3 intravenous (IV) infusions of placebo
  Interventions: Other: Placebo: Group 1 in Part B and Part C
- Group 2 in Part B and Part C (Experimental): All eligible Part B and Part C participants will receive 3 intravenous (IV) infusions of KAN-101 Dose 3
  Interventions: Drug: Group 2 in Part B and Part C
- Group 3 in Part B and Part C (Experimental): All eligible Part B and Part C participants will receive 3 intravenous (IV) infusions of KAN-101 Dose 4
  Interventions: Drug: Group 3 in Part B and Part C
- Group 4 in Part B and Part C (Experimental): All eligible Part B and Part C participants will receive 3 intravenous (IV) infusions of KAN-101 Dose 5
  Interventions: Drug: Group 4 in Part B and Part C

INTERVENTIONS:
Drug: Cohort 1 in Part A — Dose 1 KAN-101 Intravenous (IV) infusion
  Other Names: KAN-101
  Arms: Cohort 1 in Part A
Drug: Cohort 2 in Part A — Dose 2 KAN-101 Intravenous (IV) infusion
  Other Names: KAN-101
  Arms: Cohort 2 in Part A
Other: Placebo: Group 1 in Part B and Part C — Placebo Intravenous (IV) infusion
  Other Names: Placebo
  Arms: Group 1 in Part B and Part C
Drug: Group 2 in Part B and Part C — Dose 3 KAN-101 Intravenous (IV) infusion
  Other Names: KAN-101
  Arms: Group 2 in Part B and Part C
Drug: Group 3 in Part B and Part C — Dose 4 KAN-101 Intravenous (IV) infusion
  Other Names: KAN-101
  Arms: Group 3 in Part B and Part C
Drug: Group 4 in Part B and Part C — Dose 5 KAN-101 Intravenous (IV) infusion
  Other Names: KAN-101
  Arms: Group 4 in Part B and Part C

SUMMARY:
This study is to evaluate the Pharmacodynamic (PD), safety, tolerability, Pharmacokinetic (PK), and plasma biomarker response of KAN-101 in participants with Celiac Disease (CeD).

DETAILED DESCRIPTION:
The study is a 3-part, multicenter Phase 1b/2 study of KAN-101 in participants with Celiac Disease (CeD) on a gluten free diet (GFD). The 3 parts include:

* Part A - Open-label, multiple ascending dose
* Part B - Double-blind, placebo-controlled, parallel design
* Part C - Double-blind, placebo-controlled, parallel design

Part A is a Phase 1b, open-label, multiple ascending dose (MAD) study design to assess the safety, tolerability, and pharmacokinetics (PK) of KAN-101 in adult participants (18 to 70 years inclusive) with histology-confirmed CeD. Up to 12 participants who meet study inclusion/exclusion criteria will receive 1 of 2 dose levels of KAN-101. The overall study duration will be about 56 days, including up to 28 days of screening, 7 days of treatment and 21 days of follow up. There will be a gluten challenge test (GC) on Day 15.

Parts B and C are Phase 2, double-blind, placebo-controlled, parallel design study to characterize the biomarker response following GC, safety, tolerability, and PK of KAN-101 in adult participants with histology-confirmed CeD. Approximately 16 participants (4 participants per dose group) will be enrolled in Part B and 104 participants (26 participants per dose group) enrolled into Part C. Participants will be randomized 1:1:1:1 and stratified by participation in a biopsy substudy to 4 treatment groups: placebo and 3 treatment groups with KAN-101 doses based on information obtained from Part A.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of celiac disease based on histology and positive celiac serology
* HLA-DQ2.5 genotype
* Gluten-free diet for at least 12 months
* Negative or weak positive for transglutaminase IgA and negative or weak positive for DGP-IgA/IgG during screening

Exclusion Criteria:

* Refractory celiac disease
* HLA-DQ8 genotype
* Previous oral gluten challenge within 12 months
* Selective IgA deficiency
* Diagnosis of Type-1 diabetes
* Active gastrointestinal diseases
* History of dermatitis herpetiformis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of TEAEs as assessed by common terminology criteria for adverse events (CTCAE) in Part A | 28 days
  Primary endpoint in Part A. CTCAE is a scale with 5 grades to assess AE severity.
Change in magnitude of IL-2 response pre- and post-GC in peripheral blood in Part B | Baseline to Day 15
  Primary endpoint in Part B
Change in magnitude of IL-2 response pre- and post-GC in peripheral blood | 0 (pre-GC) and 4 hours post-GC on Day 15
  Primary endpoint in Part C

SECONDARY OUTCOMES:
KAN-101 plasma exposure in Part A: AUCinf | 0 (pre-dose) and up to 7 hours post dose
  PK sample collection at pre- dose and post dose timepoints in Part A.
KAN-101 plasma exposure in Part A: AUClast | 0 (pre-dose) and up to 7 hours post dose
  PK sample collection at pre- dose and post dose timepoints in Part A.
KAN-101 plasma exposure in Part A: Cmax | 0 (pre-dose) and up to 7 hours post dose
  PK sample collection at pre- dose and post dose timepoints in Part A.
KAN-101 plasma exposure in Part A: Tmax | 0 (pre-dose) and up to 7 hours post dose
  PK sample collection at pre- dose and post dose timepoints in Part A.
KAN-101 plasma exposure in Part A: t½ | 0 (pre-dose) and up to 7 hours post dose
  PK sample collection at pre- dose and post dose timepoints in Part A.
KAN-101 plasma exposure in Part B and Part C: AUCinf | 0 (pre-dose) and up to 4 hours post dose
  PK sample collection at pre- dose and post dose timepoints in Part B and Part C.
KAN-101 plasma exposure in Part B and Part C: AUClast | 0 (pre-dose) and up to 4 hours post dose
  PK sample collection at pre- dose and post dose timepoints in Part B and Part C.
KAN-101 plasma exposure in Part B and Part C: Cmax | 0 (pre-dose) and up to 4 hours post dose
  PK sample collection at pre- dose and post dose timepoints in Part B and Part C.
KAN-101 plasma exposure in Part B and Part C: Tmax | 0 (pre-dose) and up to 4 hours post dose
  PK sample collection at pre- dose and post dose timepoints in Part B and Part C.
KAN-101 plasma exposure in Part B and Part C: t½ | 0 (pre-dose) and up to 4 hours post dose
  PK sample collection at pre- dose and post dose timepoints in Part B and Part C.
Incidence and severity of TEAE as assessed by the CTCAE in Part B and Part C. | Week 52
  Secondary endpoint in Part B and Part C

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Anokion SA
Locations (36):
- United States (23):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - GCP Research, St. Petersburg, Florida
  - Agile Clinical Research Trials, Sandy Springs, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Sneeze, Wheeze & Itch Associates, LLC, Normal, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Quality Clinical Research, Omaha, Nebraska
  - Celiac Disease Center at Columbia University, New York, New York
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Aventiv Research, Inc. d/b/a Centricity Research, Columbus, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Northshore Gastroenterology Research, LLC, Westlake, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Digestive Research of Central Texas, Waco, Texas
  - Advanced Research Institute, Ogden, Utah
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
- Australia (6):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Wesley Research Institute, Auchenflower, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - St John of God Midland Public and Private Hospitals, Midland, Western Australia
- New Zealand (7):
  - PCRN Trials, Takapuna, Auckland
  - P3 Research - Tauranga, Tauranga, Bay of Plenty
  - P3 Research - Dunedin, Dunedin, Otago
  - P3 Research - Palmerston North, Paraparaumu, Wellington Region
  - Optimal Clinical Trials, Auckland
  - Waikato Hospital, Hamilton
  - P3 Research - Wellington, Wellington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murray JA, Wassaf D, Dunn K, Arora S, Winkle P, Stacey H, Cooper S, Goldstein KE, Manchanda R, Kontos S, Grebe KM. Safety and tolerability of KAN-101, a liver-targeted immune tolerance therapy, in patients with coeliac disease (ACeD): a phase 1 trial. Lancet Gastroenterol Hepatol. 2023 Aug;8(8):735-747. doi: 10.1016/S2468-1253(23)00107-3. Epub 2023 Jun 14. PMID 37329900